CLINICAL TRIAL: NCT04484779
Title: User Experience and Daily Use Patterns With the Integrated Insulin Management (IIM) System
Brief Title: A Study of an Insulin Management System in Participants With Type 1 or Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16928; F3Z-MC-IOQY (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-07-10; First posted 2020-07-24 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- IIM System (Experimental): The IIM system is comprised of an insulin lispro pen and/or an insulin glargine pen (both U-100), an investigational mobile medical application (MMA) that transmits data to cloud storage, an investigational Bluetooth Low Energy® (BLE)-paired insulin data transmission (IDT) module and a compatible commercially available BLE-paired blood glucose meter (BGM).
  Interventions: Device: IIM System; Drug: Insulin Lispro and/or Insulin Glargine

INTERVENTIONS:
Device: IIM System — IIM System
Drug: Insulin Lispro and/or Insulin Glargine — Administered subcutaneously (SC)

SUMMARY:
The purpose of this study is to investigate the user experience of an integrated insulin management system (IIM) in participants with type 1 or type 2 diabetes. The IIM system is comprised of an insulin injection pen with a data transmission module and blood glucose meter which are connected to a mobile phone application. The application will be used to record and track diabetes-data related information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed (clinically) with type 1 diabetes (T1D) for at least 1 year or type 2 diabetes (T2D) for at least 6 months.
* Using insulin injection regimen of basal/bolus or basal only for 3 months prior to screening, which includes:

  * for bolus insulin (U-100) - a rapid-acting insulin analog (glulisine, lispro, or aspart).
  * for basal insulin - degludec (U-100 or U-200), detemir (U-100), or glargine (U- 100 or U-300).
* Participants with T2D may be on ≤ 3 anti-hyperglycemic medications in addition to insulin, including alpha-glucosidase inhibitors, dipeptidyl peptidase 4 (DPP-4) inhibitors, glucagon-like peptide 1 receptor agonist (GLP-1 RA; oral or injectable), meglitinides, metformin, sodium-glucose cotransporter-2 inhibitors (SGLTi-2), sulfonylureas, or thiazolidinediones consistent with product labeling.
* Participants with T1D must be on insulin only.
* Have point-of-care hemoglobin A1c (HbA1c) value of ≤11% at screening.
* Must be able to self-inject insulin dose (basal or basal/bolus) without assistance.
* If using Continuous Glucose Monitoring or Flash Glucose Monitoring device, must agree to stop use throughout duration of trial.
* Must be able to read and speak English.
* Able and willing to use only study-provided insulin Basaglar and/or Humalog for duration of trial.
* Able and willing to follow insulin regimen specified by investigator throughout duration of trial, insulin dose may be titrated at investigator's discretion.
* Have no physical or cognitive disabilities that would, in the opinion of the investigator, preclude participant from using sponsor-provided iOS device for study activities and comply with study requirements.
* Agree not to post any personal medical data, pictures of the IIM system or information related to the study on any website or social media site (for example, Facebook, Twitter, LinkedIn, etc.).
* Have refrigeration in home for storage of insulin.
* Women of childbearing potential participating:

  * Cannot be pregnant or intend to become pregnant during the trial period
  * Cannot be breastfeeding (including the use of a breast pump)
  * Must remain abstinent or
  * Must use 1 highly effective method (less than 1% failure rate) of contraception or a combination of 2 effective methods of contraception for the entirety of the study and
  * Test negative for pregnancy based on a urine pregnancy test at the time of screening. Additional local urine pregnancy tests may be conducted for duration of trial at discretion of investigator.

Exclusion Criteria:

* If not able to take the basal insulin dose in 1 injection per day.
* Have experienced an episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within 3 months prior to screening.
* Have hypoglycemia unawareness as judged by the investigator.
* Have had 1 or more emergency room visits or hospitalization due to poor glucose control (hyperglycemia or diabetic ketoacidosis [DKA]) within 3 months prior to screening.
* History of renal transplantation, receiving renal dialysis, or diagnosed with stage IV chronic kidney disease.
* Any of the following cardiovascular conditions within 6 months prior to screening: i. acute myocardial infarction (MI) ii. cerebrovascular accident (stroke) iii. unstable angina, or iv. hospitalization due to congestive heart failure (CHF)
* Presence or history of severe congestive heart failure (New York Heart Association Class IV [CCNYHA 1994]).
* Have history of or clinical signs of liver disease (for example, acute or chronic hepatitis, or cirrhosis).
* Have active or untreated malignancy except basal cell or squamous cell skin cancer.
* Have any hypersensitivity or allergy to any of the insulins or excipients used in this trial.
* Have vision loss or vision impairment that does not allow recognition of MMA screen features.
* Have impaired dexterity which limits ability to use injection device or mobile MMA.
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have participated, within the last 30 days, in a clinical study involving an investigational product. If the previous investigational product has a long halflife, 5 half-lives or 30 days (whichever is longer) should have passed.
* Have previously completed or withdrawn from this study.
* Have previously used or are currently using an approved or investigational connected pen system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Total and Domain Specific Score of the mHealth App Usability Questionnaire (MAUQ) for Standalone mHealth Apps Used by Patients | 10 Weeks
  Total and Domain Specific Score of the MAUQ for Standalone mHealth Apps Used by Patients

SECONDARY OUTCOMES:
Overall Ease of Use of the IIM System | 10 Weeks
  Overall Ease of Use of the IIM System Assessed by the Participant Feedback Form
Likelihood of Site to Recommend the IIM System | 10 Weeks
  Likelihood of Site to Recommend the IIM System Assessed by the Site Feedback Form

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-532-0186 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Medical Investigations Inc., Little Rock, Arkansas
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No